CLINICAL TRIAL: NCT04081246
Title: Transurethral Modified En Bloc Resection For Large Bladder Tumours.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Jeremy Yuen Chun TEOH, Assistant Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CREC 2018.580-T
Record Dates: First submitted 2019-09-05; First posted 2019-09-09 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Bladder Cancer; Bladder Neoplasm; Bladder Tumor
Keywords: Bladder cancer, bladder tumour, en bloc resection
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Modified en bloc resection (Experimental): For patients undergoing modified en bloc resection, piecemeal resection of the exophytic part of the bladder tumour will be performed, followed by en bloc resection of the tumour base.
  Interventions: Device: Bipolar transurethral modified en bloc resection of bladder tumour

INTERVENTIONS:
Device: Bipolar transurethral modified en bloc resection of bladder tumour — Olympus TURis Bipolar HF-resection electrode (Model: WA22306D)

SUMMARY:
Modified en bloc resection is a hybrid technique involving piecemeal resection of the exophytic part of the bladder tumour, followed by en bloc resection of the tumour base. In this study, we shall investigate the efficacy of modified en bloc resection for patients with bladder tumours of ≥3cm in size.

DETAILED DESCRIPTION:
The biggest limiting factor of en bloc resection is the size of the bladder tumour. Resection of the bladder tumour is technically feasible, but the retrieval of specimen in one piece is restricted by the narrow size of the urethra. However, the greatest advantage of en bloc resection is to ensure complete local resection rather than the theoretical benefit of avoiding tumour re-implantation. Therefore, the concept of modified en bloc resection for large bladder tumours of ≥3cm has evolved. It is a hybrid technique involving piecemeal resection of the exophytic part of the bladder tumour, followed by en bloc resection of the tumour base. By resecting the exophytic part of the bladder tumour, the size of main tumour bulk can be reduced. By performing en bloc resection of the tumour base, the advantage of ensuring complete tumour resection beneath the submucosal plane can be preserved, and the tumour base specimen remains intact for histological assessment of the resection margins. Modified en bloc resection is a promising surgical technique which can potentially ensure complete tumour resection, reduce the need of second-look transurethral resection, and improve the oncological control of non-muscle-invasive bladder cancer in long run. It may also ensure proper staging of muscle-invasive bladder cancer at the first surgery, thus avoiding the need of second-look transurethral resection in under-staged patients.

In this study, we shall evaluate the efficacy of modified en bloc resection for patients with bladder tumours of ≥3cm. All patients will have MRI before modified en bloc resection. All patients with non-muscle-invasive bladder cancer will be offered second-look transurethral resection in 2-6 weeks' time. All patients with muscle-invasive bladder cancer but not distant metastasis will be offered radical cystectomy, pelvic lymphadenectomy and urinary diversion; for those who refuse or who are considered unfit for radical surgery, second-look transurethral resection will be offered. All patients will have a second MRI before the second surgery. The modified en bloc resection specimen results will be compared with the final pathology results in the second surgery. The presence of any residual or upstaging of disease will be determined. The results of the two sets of MRI will also be compared with the final pathology results. The accuracy of MRI in the evaluation of bladder cancer will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80 years old with informed consent
* Bladder tumours with maximal dimension of ≥ 3cm

Exclusion Criteria:

* Bladder tumour detected during intravesical Bacillus Calmette-Guerin therapy (These patients warrant more aggressive treatment, i.e. radical cystectomy)
* Estimated glomerular filtration rate of <60mL/min.
* Presence of clinically significant cardiovascular disease (History of acute myocardial infarction, presence of uncontrolled angina within 3 months before screening, New York Heart Association Class III or IV congestive heart failure, presence of ventricular arrhythmias, or presence of second-degree or third-degree heart block)
* Presence of GOLD Stage III or IV chronic obstructive pulmonary disease
* History of bleeding disorder or use of anti-coagulant
* Presence of other active malignancy
* ECOG performance status ≥ 2 (Ambulatory and capable of all self care but unable to carry our any work activities. Confined to bed or chair less than 50% of waking hours)
* Pregnancy
* Presence of metallic foreign body or implant which is not MRI compatible
* Known history of claustrophobia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-09-07 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Composite outcome on the rate of complete resection for non-muscle-invasive bladder cancer and proper staging for muscle-invasive bladder cancer | Seven weeks after the experimental operation
  Complete resection for non-muscle-invasive bladder cancer is defined as the absence of any malignancy upon second-look transurethral resection surgery, in patients who have non-muscle-invasive bladder cancer upon the first modified en bloc resection. Proper staging for muscle-invasive bladder cancer is defined as the detection of muscle-invasive bladder cancer upon the first modified en bloc resection, in all patients who have a definitive histological diagnosis of muscle-invasive bladder cancer upon modified en bloc resection or second-look transurethral resection surgery. Second look transurethral resection surgery is expected to perform within six weeks after the experimental operation and one more week is allowed for histological assessment of the second look transurethral resection specimen.

SECONDARY OUTCOMES:
Proper staging rate for non-muscle-invasive bladder cancer | Seven weeks after the experimental operation
  The proper staging rate for non-muscle-invasive bladder cancer is defined as the absence of any upstaging of the T-stage upon second-look transurethral resection surgery, in patients who have non-muscle-invasive bladder cancer upon the first modified en bloc resection. Second look transurethral resection surgery is expected to perform within six weeks after the experimental operation and one more week is allowed for histological assessment of the second look transurethral resection specimen.
Complete resection rate for muscle-invasive bladder cancer | Seven weeks after the experimental operation
  The complete resection rate for muscle-invasive bladder cancer is defined as the absence of any malignancy upon second-look transurethral resection surgery or radical surgery, in patients who have muscle-invasive bladder cancer upon the first modified en bloc resection. Second look transurethral resection surgery or radical surgery are expected to perform within six weeks after the experimental operation and one more week is allowed for histological assessment of the second look transurethral resection specimen.
Successful modified en bloc resection rate | Immediately post-operative
  Techical success rate of modified en bloc resection
Negative circumferential resection margin rate | One week after the experimental operation
  Rate of negative circumferential resection margin of the modified en bloc resection pathological specimen
Negative deep resection margin rate | One week after the experimental operation
  Rate of negative deep resection margin of the modified en bloc resection pathological specimen
Detrusor muscle sampling rate | One week after the experimental operation
  Rate of presence of detrusor muscle in the modified en bloc resection pathological specimen
Occurrence of obturator reflex | Intra-operative
  Number of participants with obturator reflex encountered by the operating surgeon during the modified en bloc resection operation
Operative time | Immediately post-operative
  Duration of operation
Rate of mitomycin C instillation | Immediately post-operative
  One day after the experimental operation
Duration of bladder irrigation | Three days after the experimental operation.
  Duration of bladder irrigation. Patients undergoing transurethral resection surgery have an average hospital stay of three days. Bladder irrigation is always stopped before the patient is discharged
Duration of urethral catheterisation | Three days after the experimental operation
  Duration of urethral catheterisation. Patients undergoing transurethral resection surgery have an average hospital stay of three days. Urethral catheter is often removed before the patient is discharged
Hospital stay | Three days after the experimental operation
  Patients undergoing transurethral resection surgery have an average hospital stay of three days.
30-day complications | Thirty days after the experimental surgery
  Complications which occur within 30 days after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy YC Teoh, MBBS, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ukai R, Kawashita E, Ikeda H. A new technique for transurethral resection of superficial bladder tumor in 1 piece. J Urol. 2000 Mar;163(3):878-9. PMID 10687997
- [Background] Divrik RT, Sahin AF, Yildirim U, Altok M, Zorlu F. Impact of routine second transurethral resection on the long-term outcome of patients with newly diagnosed pT1 urothelial carcinoma with respect to recurrence, progression rate, and disease-specific survival: a prospective randomised clinical trial. Eur Urol. 2010 Aug;58(2):185-90. doi: 10.1016/j.eururo.2010.03.007. Epub 2010 Mar 19. PMID 20303646
- [Background] Babjuk M, Bohle A, Burger M, Capoun O, Cohen D, Comperat EM, Hernandez V, Kaasinen E, Palou J, Roupret M, van Rhijn BWG, Shariat SF, Soukup V, Sylvester RJ, Zigeuner R. EAU Guidelines on Non-Muscle-invasive Urothelial Carcinoma of the Bladder: Update 2016. Eur Urol. 2017 Mar;71(3):447-461. doi: 10.1016/j.eururo.2016.05.041. Epub 2016 Jun 17. PMID 27324428
- [Background] Stein JP, Lieskovsky G, Cote R, Groshen S, Feng AC, Boyd S, Skinner E, Bochner B, Thangathurai D, Mikhail M, Raghavan D, Skinner DG. Radical cystectomy in the treatment of invasive bladder cancer: long-term results in 1,054 patients. J Clin Oncol. 2001 Feb 1;19(3):666-75. doi: 10.1200/JCO.2001.19.3.666. PMID 11157016